CLINICAL TRIAL: NCT05849428
Title: Blood Glucose Differences Between Left Arm and Right Arm in Patients With Type 1 or Type 2 Diabetes Using a Continuous Glucose Monitor
Brief Title: Blood Glucose Differences Using CGMs Between the Left and Right Arm in Patients With Diabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of the Pacific (Other)
Responsible Party: Principal Investigator, Sachin Shah, Professor of Pharmacy, University of the Pacific
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRB2023-25
Record Dates: First submitted 2023-04-28; First posted 2023-05-08 (Actual); Last update posted 2023-05-08 (Actual); Status verified 2023-04

CONDITIONS: Type 1 Diabetes; Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2 | interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Measuring Arm (Other): Participants will wear 2 Freestyle Libre 3 sensors on each arm, 1 on the left and 1 on the right for 2 consecutive weeks (total of 14 days).
  Interventions: Device: Freestyle Libre 3

INTERVENTIONS:
Device: Freestyle Libre 3 — Freestyle Libre 3 consists of a sensor that is applied to the back of the upper arm. The sensor is a penny-sized flexible filament placed beneath the skin surface to measure interstitial fluid. This sensor is applied utilizing a sensor applicator provided in the packaging. The sensor will continuously read interstitial glucose readings every minute and syncs with the Freestyle View app. At the completion of the study, the sensor is discarded per protocol.
  Other Names: Continuous Glucose Monitoring (CGM) device

SUMMARY:
There are multiple CGMs that are FDA approved. However, there are few studies looking at the variability of measurements between the left and right arm, and none looking at this effect in diabetic patients. This study may identify if glucose differences exist in the left and right arm in patients with Type 1 or Type 2 Diabetes. Furthermore, it may point to future directions for research to standardize methods of glucose measurement such as consistently measuring on only one side of the body.

DETAILED DESCRIPTION:
The goal of this clinical trial is to determine the time-matched difference in glucose levels between the left arm and right arm in patients with Type 1 or Type 2 diabetes. The main objective aims to answer:

• Is there a difference in time-matched controlled glucose monitoring (CGM) - derived blood glucose between left and right arm in patients with Type 1 or Type 2 diabetes in target range (<70 mg/dL; 70-180 mg/dL; >180 mg/dL)?

Participants will wear two Freestyle Libre 3 sensors, 1 on the left and 1 on the right arm, continuously for 2 weeks. Participants will need to download the Freestyle Libre 3 app on two separate mobile devices and connect the sensors with Freestyle Libre View accounts provided by the study team. The study team will collect and compare the data between the left and right arm for further analysis.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18-65 years of age
* Diagnosed with Type 1 or Type 2 Diabetes
* Willing to wear CGMs for 2 weeks on both arms
* Willing to attend 3 virtual calls meetings over the course of the trial
* Have active health insurance
* Willing to refrain from any heat therapy for the duration of the study
* Willing to refrain from consuming ascorbic acid and salicylic acid for the duration of the study due to known interaction with CGMs
* Have access to 2 compatible mobile devices for the Freestyle Libre 3 CGMs
* Not currently using any Freestyle Libre CGM
* Willing to provide HbA1c readings within 3 months of the trial
* Have a baseline HbA1c equal or above 6.5

Exclusion Criteria:

* Any active dermatologic condition on the upper arms
* Implanted medical devices including another continuous glucose monitoring device (i.e.

pacemaker)

* Critically ill or dialysis patients
* Planned magnetic resonance imaging screening, computed tomography scan, X-ray imaging or high-frequency electrical heat treatment during study period
* Current systemic infections
* Subjects who are unable to fully understand the study or consent process will not be included in the study due to the lack of a qualified medical translator
* Refusal to sign the informed consent document
* Pregnant, planned pregnancy during study period, or currently breast-feeding
* Fear of needles to the point where patients cannot self-administer the sensors
* History of allergic reactions or hypersensitivity from adhesives

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-05 (Estimated); Primary Completion 2023-06 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Time-matched CGM-derived blood glucose differences between left arm and right arm in patients with Type 1 or Type 2 Diabetes below target range (<70 mg/dL). | 14 days
  Data gathered from the CGM device will be sync'd with the Freestyle View app and made available to the study team for analysis below the target range (<70 mg/dL).

SECONDARY OUTCOMES:
Time-matched CGM-derived blood glucose differences between left arm and right arm in patients in target range (70-180 mg/dL). | 14 days
  Data gathered from the CGM device will be sync'd with the Freestyle View app and made available to the study team for analysis at the target range (70-180 mg/dL).
Time-matched CGM-derived blood glucose differences between left arm and right arm in patients above target range (>180 mg/dL). | 14 days
  Data gathered from the CGM device will be sync'd with the Freestyle View app and made available to the study team for analysis at the target range (>180180 mg/dL).

CONTACTS AND LOCATIONS:
Locations (1):
- University of the Pacific, Stockton, California, United States

REFERENCES:
- [Background] Juvenile Diabetes Research Foundation Continuous Glucose Monitoring Study Group; Beck RW, Hirsch IB, Laffel L, Tamborlane WV, Bode BW, Buckingham B, Chase P, Clemons R, Fiallo-Scharer R, Fox LA, Gilliam LK, Huang ES, Kollman C, Kowalski AJ, Lawrence JM, Lee J, Mauras N, O'Grady M, Ruedy KJ, Tansey M, Tsalikian E, Weinzimer SA, Wilson DM, Wolpert H, Wysocki T, Xing D. The effect of continuous glucose monitoring in well-controlled type 1 diabetes. Diabetes Care. 2009 Aug;32(8):1378-83. doi: 10.2337/dc09-0108. Epub 2009 May 8. PMID 19429875
- [Background] Siegmund T, Heinemann L, Kolassa R, Thomas A. Discrepancies Between Blood Glucose and Interstitial Glucose-Technological Artifacts or Physiology: Implications for Selection of the Appropriate Therapeutic Target. J Diabetes Sci Technol. 2017 Jul;11(4):766-772. doi: 10.1177/1932296817699637. Epub 2017 Mar 21. PMID 28322063
- [Background] Shapiro AR. Nonadjunctive Use of Continuous Glucose Monitors for Insulin Dosing: Is It Safe? J Diabetes Sci Technol. 2017 Jul;11(4):833-838. doi: 10.1177/1932296816688303. Epub 2017 Mar 1. PMID 28540756
- [Background] American Diabetes Association. 6. Glycemic Targets: Standards of Medical Care in Diabetes-2020. Diabetes Care. 2020 Jan;43(Suppl 1):S66-S76. doi: 10.2337/dc20-S006. PMID 31862749
- [Background] Vigersky RA, McMahon C. The Relationship of Hemoglobin A1C to Time-in-Range in Patients with Diabetes. Diabetes Technol Ther. 2019 Feb;21(2):81-85. doi: 10.1089/dia.2018.0310. Epub 2018 Dec 21. PMID 30575414
- See also: 957-P: Differences in Glucose Level between Left Arm and Right Arm Using Continuous Glucose Monitors — https://doi.org/10.2337/db19-957-P
- See also: FreeStyle Libre 2-Best Glucose Monitor For Kids - Coming Soon for Patients 4+. Continuous Glucose Monitoring System. — https://www.freestyle.abbott/us-en/products/freestyle-libre-2.html